CLINICAL TRIAL: NCT07382726
Title: Combination Of Izalontamab Brengitecan And Adagrasib In Advanced KRAS G12Ci-Refractory Non-Small Cell Lung Cancer - The IZA-A Trial
Brief Title: Phase 1 Study Of Izalontamab Brengitecan + Adagrasib In NSCLC - The IZA-A Trial
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1306; NCI-2026-00662 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — adagrasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combo Treatment with Izalontamab Brengitecan (IV) + Adagrasib (PO) Q3W (Experimental): Adagrasib will be administered at 400mg PO BID continuously. Iza-bren will be administered IV on Day 1 and Day 8 (+3 days) in a 21-day cycle.
  Interventions: Drug: Adagrasib; Drug: Iza-bren

INTERVENTIONS:
Drug: Adagrasib — Given by mouth
  Other Names: Krazati
Drug: Iza-bren — Given by IV

SUMMARY:
This research is being done to test a combination of two drugs, Izalontamab Brengitecan (iza-bren) and Adagrasib, in patients with advanced KRAS G12C-mutant NSCLC that hasn't responded to other treatments. The purpose is to see if this combination works better than existing treatments for people whose cancer keeps growing despite KRAS G12C inhibitors.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the safety and tolerability of iza-bren in combination with adagrasib for treatment of KRAS G12C-mutant NSCLC patients that progressed on KRAS G12C inhibitors.

Secondary Objectives:

* To evaluate the preliminary efficacy of iza-bren in combination with adagrasib for treatment of KRAS G12C-mutant NSCLC patients that progressed on KRAS G12C inhibitors.
* To evaluate the pharmacokinetics of iza-bren upon combination treatment with adagrasib.
* To evaluate immunogenicity against iza-bren upon combination treatment with adagrasib.
* To evaluate the incidence of anti-drug antibody (ADA) formation to Iza-bren when it is administered in combination with adagrasib, and to assess the potential effect of ADA on PK, PD and safety.
* To evaluate EGFR and HER3 tumor expression as determinants of clinical outcomes to study regimen.
* To evaluate circulating tumor DNA (ctDNA) as a determinant of clinical outcome to study regimen.
* To evaluate mechanisms of resistance to study regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of NSCLC or NSCLC predominant histology.
* Patients must have a diagnosis of metastatic or locally advanced NSCLC not amenable to curative therapy
* Tumor must harbor a KRAS G12C mutation. Testing available through multigene NGS panels performed in the Molecular Diagnostics Laboratory in UT MD Anderson Cancer Center and can be performed using either tissue or blood assays. Use of standard of care (SOC) results are allowed to meet this requirement.
* Patients must have progressed on a prior KRAS G12C inhibitor as monotherapy or as combination therapy.
* Patients must have received at least one prior line of therapy and up to 3 prior lines of therapy.
* Patients must have measurable disease per RECIST v1.1.
* Age ≥18 years - no dosing or adverse event data are currently available on the use of izabren and adagrasib in patients <18 years of age; children are excluded from this study.
* ECOG performance status 0 - 1.
* Most recent prior systemic therapy (e.g., chemotherapy, immunotherapy or, investigational agent) discontinued at least 2 weeks before first dose date.
* Most recent radiation treatment discontinued at least 1 week prior to first dose date (includes brain radiation).
* Patients must have adequate organ and marrow function as defined below:

Hemoglobin ≥9.0g/dL Absolute neutrophil count ≥1,500/mcL Platelets ≥100,000/mcL Total bilirubin ≤ institutional upper limit of normal (ULN) (if associated with liver metastases or Gilbert's disease, ≤ 3 x ULN) AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN (if associated with liver metastases, ≤ 5 x ULN) Creatinine ≤ 1.5 mg/dL or CrCl ≥ 45 mL/min (calculated using a validated prediction equation - e.g., Cockcroft-Gault, MDRD, or 24-hour urine CrCl)

* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable.
* Patients with a history of hepatitis C virus (HCV) infection must have documentation of undetectable HCV viral load.
* Patients with treated brain metastases are eligible if patients are neurologically stable for at least 1 week prior to the first dose of study treatment without the use of corticosteroids or are on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent).
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* Because adagrasib and iza-bren are known to be teratogenic, women of child-bearing potential (WCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 4 (men) and 7 (WCBP) months after completion of study treatment administration. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients less than 55 years of age unless the patient presents with an applicable exclusionary factor which may be one of the following:

  * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
  * History of hysterectomy or bilateral salpingo-oophorectomy.
  * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
  * History of bilateral tubal ligation or another surgical sterilization procedure.
* Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 4 months after completion of study treatment administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) except for alopecia and parameters superseded by other eligibility criteria [e.g., laboratory parameters]).
* Patients who are receiving any other investigational agents.
* Patients with active untreated brain metastases or carcinomatous meningitis.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to adagrasib and iza-bren.
* Patients with prior history of pneumonitis or interstitial lung disease. Patients with prior history of radiation pneumonitis which was asymptomatic or resolved with steroid treatment, and without evidence of clinically active radiation pneumonitis are eligible.
* Human immunodeficiency virus (HIV)-infected patients. Those on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and actively breastfeeding woman due to concerns for teratogenicity and infant toxicity.
* Major surgery within 4 weeks prior to first dose of study treatment.
* History of intestinal disease or major gastric surgery likely to alter absorption of study treatment or inability to swallow oral medications.
* Prolonged QTc interval (>470 milliseconds for women and >450 milliseconds for men), or immediate family or medical history of congenital Long QT Syndrome.
* History of stroke or transient ischemic attack within 6 months prior to first dose of study treatment.
* History of unstable angina, myocardial infarction, and symptomatic atrial fibrillation within 6 months prior to first dose of study treatment.
* Any serious illness, uncontrolled inter-current illness, psychiatric illness, active or uncontrolled infection, or other medical history, including laboratory results, which, in the Investigator's opinion, would be likely to interfere with the patient's participation in the study, or with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-12-24 (Estimated); Study Completion 2029-12-24 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo V Negrao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org